CLINICAL TRIAL: NCT00443118
Title: NEWBORN VENTILATION IN THE DELIVERY ROOM: CAN IT BE IMPROVED WITH A T-PIECE RESUSCITATOR? Multicenter Cross-over Cluster Randomized Controlled Trial
Brief Title: Newborn Ventilation in the Delivery Room: Could it be Improved With a T-piece Resuscitator?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Edgardo Szyld (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Edgardo Szyld, Principal Investigator, Fundacion para la Salud Materno Infantil
Organization: Fundacion para la Salud Materno Infantil (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fundasamin 102; NCT01126489 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Resuscitation
Keywords: Bag and mask; Neopuff; Resuscitation; Newborn; Intubation; devices; PEEP
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neopuff TM with PEEP (Active Comparator): Newborns ventilated for neonatal resuscitation using Neopuff TM with PEEP
  Interventions: Device: T-piece resuscitator Neopuff TM
- Self Inflating Bag with PEEP (Active Comparator): Newborns ventilated for neonatal resuscitation using Self Inflating Bag with PEEP valve attached
  Interventions: Device: Self Inflating Bag with PEEP
- Self Inflating Bag without PEEP (Active Comparator): Newborns ventilated for neonatal resuscitationusing Self Inflating Bag without PEEP valve attached
  Interventions: Device: Self Inflating Bag without PEEP

INTERVENTIONS:
Device: T-piece resuscitator Neopuff TM — Positive pressure ventilation will be performed with Neopuff® with face mask. For this study, an initial PIP 25 cm H2O and a 5 cm H2O PEEP will be used for resuscitation according to protocol.
  Arms: Neopuff TM with PEEP
Device: Self Inflating Bag with PEEP — Positive pressure ventilation will be performed with Self Inflating Bag with PEEP with face mask. For this study, an initial PIP 25 cm H2O and a 5 cm H2O PEEP will be used for resuscitation according to protocol.
  Other Names: Ambu
  Arms: Self Inflating Bag with PEEP
Device: Self Inflating Bag without PEEP — Positive pressure ventilation will be performed with Self Inflating Bag without PEEP with face mask. For this study, an initial PIP 25 cm H2O and a 5 cm H2O PEEP will be used for resuscitation according to protocol.
  Other Names: Ambu
  Arms: Self Inflating Bag without PEEP

SUMMARY:
A multicenter cross-over cluster randomized controlled trial protocol study in newborn infants ≥ 26 weeks gestational age requiring assisted ventilation (positive pressure ventilation [PPV]) for resuscitation in the delivery room comparing a T-piece resuscitator device versus resuscitation bag.

DETAILED DESCRIPTION:
Design: A multicenter cross-over cluster randomized controlled trial. Our hypothesis is based on the assumption that ventilating depressed newborns with a T-piece resuscitator will be more effective than SIB by increasing the proportion of resuscitated newborns with heart rate (HR) ≥ 100 beats per minute (bpm) at two minutes of life as a proxy for successful resuscitation.

Population: Newborn infants ≥ 26 weeks gestational age requiring assisted ventilation (PPV) for resuscitation in the delivery room.

(need for assisted ventilation at positive pressure: Heart Rate [HR] < 100 beats per minute [bpm], apnea, gasping, cyanosis and/or hypotonia)

Intervention: PPV will be performed with a T-piece resuscitator (Neopuff® group) with positive end expiratory pressure.

Control: PPV will be performed with a self inflating bag (SIB group) with and without PEEP.

Both devices will be used with face masks, and a peak inspiratory pressure (PIP) of 25 cm H2O will be used to begin ventilation with PEEP of 0 cm H2O in the subgroup without PEEP valve, 5 cm H2O in the subgroup with PEEP valve in the SIB group, and 5 cm H2O in the Neopuff® group.

Objective: To compare the effectiveness of both instruments in reaching a heart rate of ≥ 100 bpm in depressed newborns of ≥ 26 weeks' gestational age (GA) after the initiation of positive pressure ventilation (PPV) with face mask.

Primary Outcome: Proportion of newborns with HR ≥ 100 bpm at 2 minutes of life.

Type of Comparison: Which of the two devices Neopuff TM or Self Inflating Bag (NP/SIB)will be more effective for ventilation of the newborn, by increasing the proportion of resuscitated newborns with heart rate (HR) ≥ 100 beats per minute (bpm) at two minutes of life as a proxy for successful resuscitation.

ELIGIBILITY:
Inclusion criteria:

Live-born infants of ≥ 26 weeks' GA with HR < 100 bpm requiring resuscitation with positive pressure ventilation with mask in the delivery room according to the current AAP/AHA recommendations

Exclusion Criteria:

Infants requiring intubation from birth. Newborns of < 26 weeks´ GA. Newborns presenting major congenital malformations. Multiple births. Problems (difficulty or malfunctioning) with the device assigned.

Max Age: 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1032 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Szyld, MD, Principal Investigator — Fundasamin; Adriana Aguilar, MD, Study Director — Hospital Paroissien; Waldemar Carlo, MD, Study Chair — University of Alabama at Birmingham; Nestor Vain, MD, Study Director — Sanatorio de la Trinidad; Luis Prudent, MD, Study Director — Sanatorio Otamendi
Locations (11):
- United States (2):
  - Carol Jo Vecchie Women and Children's Center at St. John's Hospital, Springfield, Illinois
  - Cleveland Clinic, Cleveland, Ohio
- Argentina (4):
  - Sanatorio de los Arcos, Ciudad de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Misericordia, Córdoba
  - Nuevo Hospital El Milagro de Salta, Salta
- Chile (3):
  - Hospital Clínico de la Pontificia Universidad Católica de Chile, Santiago
  - Hospital Dr. Hernán Henriquez Aravena, Temuco
  - Hospital Dr. Gustavo Fricke, Viña del Mar
- Azienda Ospedaliera Padova, Padua, Veneto, Italy
- Instituto Nacional Materno Perinatal (INMP) de Perú, Lima, Peru

REFERENCES:
- [Derived] Szyld E, Aguilar A, Musante GA, Vain N, Prudent L, Fabres J, Carlo WA; Delivery Room Ventilation Devices Trial Group. Comparison of devices for newborn ventilation in the delivery room. J Pediatr. 2014 Aug;165(2):234-239.e3. doi: 10.1016/j.jpeds.2014.02.035. Epub 2014 Mar 29. PMID 24690329
- See also: this paper was published on The Journal of Pediatrics — http://www.ncbi.nlm.nih.gov/pubmed/24690329

RESULTS

PARTICIPANT FLOW:
Groups:
- T-Piece: Subjects assigned to be resuscitated with T-Piece
- SIB - With PEEP Valve: Subjects allocated to SIB with a PEEP valve attached
- SIB-Without PEEP Valve: Self inflating bag without PEEP valve
Period: Overall Study
Arm/Group | T-Piece | SIB - With PEEP Valve | SIB-Without PEEP Valve
Started | 515 | 291 | 226
Completed | 511 | 290 | 226
Not Completed | 4 | 1 | 0
Not completed — unknown primary outcome | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Self Inflating Bag With PEEP: Subjects allocated to Self Inflating Bag with PEEP
- Self Inflating Bag Without PEEP: Subjects allocated to Self Inflating Bag without PEEP
- Total: Total of all reporting groups
Arm/Group | T-Piece | Self Inflating Bag With PEEP | Self Inflating Bag Without PEEP | Total
Number analyzed (Participants) | 511 | 290 | 226 | 1027
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age. As the subjects are all newborns, the baseline important data includes Maternal data
  years | 28 (7) | 28 (7) | 27 (7) | 28 (7)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age of enrolled infants
  weeks | 36 (4.1) | 35 (5) | 37 (4) | 36 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 117 | 101 | 426
  Male | 303 | 173 | 125 | 601
previous deliveries [Number; unit: number of participants]
  primiparous | 220 | 137 | 106 | 463
  multiparous | 291 | 153 | 120 | 564
ANTENATAL STEROIDS [Number; unit: participants]
  YES | 142 | 84 | 72 | 298
  NO | 369 | 206 | 154 | 729

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Infants With a HR ≥ 100 Bpm at 2 Minutes of Life.
Time Frame: 2 minutes of life
Population: The analysis was performed by intention to treat
Measure: Number; unit: percentage of participants
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to SIB with PEEP valve attached
- SIB-Without PEEP Valve: Subjects allocated to SIB-Without PEEP valve attached
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
percentage of participants | 93.7 | 88 | 93

2. Secondary Outcome: Time the Newborn Takes to Reach a HR > 100 Bpm
Time Frame: 2 minutes of life
Measure: Mean (Inter-Quartile Range); unit: minutes
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to Self Inflating Bag with PEEP valve
- SIB-Without PEEP Valve: Subjects allocated to Self Inflating Bag withouth a PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
minutes | 1 [0.5 to 1.6] | 1 [0.5 to 1.8] | 1 [0.5 to 1.9]

3. Secondary Outcome: • SpO2 Value at 2 Minutes of Life.
Time Frame: 2 minutes of life
Population: the pulse-oximeter was reliable at 2 minutes in 69% of the cases in both groups.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to be ventilated using a Self Inlfating Bag with PEEP valve
- SIB-Without PEEP Valve: Sujects allocated to be ventilated with Self Inflating Bag Without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 350 | 199 | 155
percentage of oxygen saturation | 82 (14) | 80 (20) | 77 (16)

4. Secondary Outcome: • Proportion of Eligible Newborns Who Entered the Study and Who Were Intubated After Failure of PPV With Mask.
Time Frame: after 2 minutes of life
Measure: Number; unit: percentage of participants
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to Self Inflating Bag with a PEEP valve attached
- SIB-Without PEEP Valve: Subjects allocated to Self Inflating Bag without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
percentage of participants | 17 | 28 | 23

5. Secondary Outcome: • Need for Chest Compression and/or Medications
Time Frame: after 2 minutes of life
Measure: Number; unit: participants
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to SIB with PEEP valve
- SIB-Without PEEP Valve: Subjects Allocated to SIB without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants | 8 | 11 | 6

6. Secondary Outcome: Apgar Scores at 1 and 5 Minutes
Description: categorized Apgar score 1 min <=3 and categorized Apgar score 5 min <=5 The Apgar score is applied routinely by nurses and neonatologists to describe how vigorous the baby is at birth, it ranges from 0 to 10, with higher scores representing better outcomes.
Time Frame: 1-5 minutes of life
Measure: Number; unit: participants
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants
  apgar score 1 min <=3 | 153 | 111 | 66
  apgar score 5 min <=5 | 30 | 24 | 23

7. Secondary Outcome: • Incidence of Neonatal Encephalopathy During First Week of Life (Classified by Sarnat)
Time Frame: first week of life
Measure: Number; unit: participants
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants | 21 | 21 | 7

8. Secondary Outcome: • Incidence of Air Leaks
Description: included pneumothorax and Pneumomediastinum
Time Frame: after birth and during hospitalization up to four weeks
Measure: Number; unit: participants
Groups:
- SIB-Without PEEP Valve: Subjects allocated to SIB-Without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants | 13 | 6 | 2

9. Secondary Outcome: • Use of Oxygen Treatment Beyond the Delivery Room
Time Frame: during hospitalization
Measure: Number; unit: participants/
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants/ | 208 | 126 | 96

10. Secondary Outcome: Days on Oxygen
Time Frame: after birth and during hospitalization up to four weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
days | 13.8 (17) | 23 (27) | 23 (22)

11. Secondary Outcome: • Need for Mechanical Ventilation or CPAP
Time Frame: during hospitalization
Measure: Number; unit: participants
Groups:
- SIB-Without PEEP Valve: subjects allocate to SIB Without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
participants | 116 | 104 | 43

12. Secondary Outcome: Days on Mechanical Ventilation
Time Frame: after delivery and before four weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- SIB - Self Inflating Bag With PEEP Valve: Subjects allocated to Without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
days | 5.0 (7.6) | 7 (11) | 12 (17)

13. Secondary Outcome: Days on CPAP
Time Frame: after birth and during hospitalization up to four weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- SIB-Without PEEP Valve: Subjects allocated to be resuscitated with Self Inflating Bag Without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP Valve | SIB-Without PEEP Valve
Number analyzed (Participants) | 511 | 290 | 226
days | 7.83 (11.3) | 9.6 (11.5) | 5.2 (6.5)

14. Secondary Outcome: • Incidence of Intracranial Hemorrhage Grades 3-4 for Preterm Newborns <32 Weeks
Description: Incidence of intracranial hemorrhage grades 3-4 for preterm newborns <32 weeks by ultrasound evaluation
Time Frame: 1 day of life and 30 days after birth
Population: this is an analyisis among the subgroup of subjects <32 weeks GA. this is the population at risk of this outcome. It extremely unusual intracranial hemorrhage over 32 weeks GA.
Measure: Count of Participants; unit: Participants
Arm/Group | Neopuff TM With PEEP | Self Inflating Bag With PEEP | Self Inflating Bag Without PEEP
Number analyzed (Participants) | 90 | 73 | 34
Participants | 10 | 1 | 3

ADVERSE EVENTS:
Groups:
- SIB - Self Inflating Bag With PEEP: Subjects allocated to be ventilated with Self Inflating Bag with PEEP valve
- SIB Without PEEP: Subjects allocated to be ventilated with Self Inflating Bag without PEEP valve
Arm/Group | T-Piece | SIB - Self Inflating Bag With PEEP | SIB Without PEEP
Serious Adverse Events (participants affected / at risk) | 11/511 | 8/290 | 7/226
Other Adverse Events (participants affected / at risk) | 21/511 | 25/290 | 19/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Piece (N=511) | SIB - Self Inflating Bag With PEEP (N=290) | SIB Without PEEP (N=226)
mortality (General disorders) | 11 (11) | 8 (8) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Piece (N=511) | SIB - Self Inflating Bag With PEEP (N=290) | SIB Without PEEP (N=226)
bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 25 (25) | 19 (19) — BPD defined as need for oxygen at 36 weeks GA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No